CLINICAL TRIAL: NCT05356702
Title: Low-cost Detection of Dementia Using Electronic Health Records Data: Validation and Testing of the eRADAR Algorithm in a Pragmatic, Patient-centered Trial.
Brief Title: The Brain Health Study: A Pragmatic, Patient-Centered Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1R01AG067427 (NIH)
Record Dates: First submitted 2022-04-27; First posted 2022-05-02 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Dementia; Alzheimer Disease
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain Health Intervention (Experimental): * Calculate eRADAR scores using EHR data to identify eligible individuals
  * Invite eligible individuals for brain health assessment visit
  * Enter results of brain health assessment visit into EHR
  * Provide summary of results and recommended next steps to the Primary Care Physician and participant
  Interventions: Other: Brain Health Assessment
- Usual care (No Intervention): Individuals who meet eligibility criteria will receive usual care.

INTERVENTIONS:
Other: Brain Health Assessment — Research interventionists, who will be trained and licensed health practitioners (e.g., social workers), will ask participants about changes in memory or thinking and daily function, screen for depression, and administer a standard cognitive screening test. They will use a standardized note template to document results in the participant's EHR. Research interventionists will notify participants and PCPs if follow-up is recommended.
  Arms: Brain Health Intervention

SUMMARY:
The eRADAR Brain Health Study seeks to refine and test a novel, low-cost strategy for increasing dementia detection within primary care.

DETAILED DESCRIPTION:
eRADAR stands for "electronic health record (EHR) Risk of Alzheimer's and Dementia Assessment Rule." It is a low-cost tool or algorithm that uses readily available EHR data elements to identify high-risk patients. We will conduct a pragmatic randomized controlled trial to assess the impact of implementing eRADAR as part of a supported outreach process on dementia detection rates. We will also explore the impact of eRADAR implementation on healthcare utilization and patient experience.

ELIGIBILITY:
Inclusion Criteria:

* No prior diagnosis of dementia (defined from EHR diagnosis codes) and not receiving medications for dementia
* Active patient at participating clinic
* Adequate data to calculate eRADAR score

Exclusion Criteria:

- Currently receiving hospice care

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 3417 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
New dementia diagnoses | 12 months after index date
  Rate of new dementia diagnoses identified from the electronic health record (EHR) using a prespecified set of ICD-10 codes

SECONDARY OUTCOMES:
Healthcare utilization | 6 months after index date
  Number of primary care visits, laboratory tests performed, neuroimaging tests, and specialty visits or referrals, defined from EHR data
Dementia medications | 6 months after index date
  Percent of participants who receive new medications for dementia, defined from medication orders or dispensings in the electronic health record
Urgent care/emergency department visits | 1 year after index date
  Number of urgent care and emergency department visits
Hospitalizations | 1 year after index date
  Number of inpatient stays
Clinic "no shows" | 1 year after index date
  Number of scheduled visits missed
Medication adherence | 1 year after index date
  Proportion of days covered
New dementia diagnoses (secondary definitions) | 6 months after index date; 18 months after index date
  Dementia diagnosis rate in different time periods than for primary outcome, defined from EHR data
New diagnoses of mild cognitive impairment | 12 months after index date
  Rate of new diagnoses of mild cognitive impairment following the intervention, defined from EHR data
Rate of accepting brain health visit | 3 months after invitation mailed
  Proportion of people offered a brain health visit who accept and attend the visit
Positive predictive value of eRADAR algorithm | 12 months after index date
  Proportion of people with a high risk eRADAR Score who attend a brain health visit who are diagnosed with dementia

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Dublin, MD, PhD, Principal Investigator — KP Washington Health Research Institute; Deborah E. Barnes, PhD, Principal Investigator — University of California, San Francisco
Locations (5):
- United States (5):
  - Kaiser Permanente Burien Medical Center, Burien, Washington
  - Kaiser Permanente Kent Medical Center, Kent, Washington
  - Kaiser Permanente Renton Medical Center, Renton, Washington
  - Kaiser Permanente, Capitol Hill, Seattle, Washington
  - Kaiser Permanente Northgate Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
This Individual Participant Data (IPD) plan applies to all quantitative study data, such as data collected specifically for the study and those derived from electronic health records (EHR), as well as the data collected via planned study surveys, which include only short qualitative free-text fields. We do not plan to share transcripts from in-depth qualitative interviews or recorded study assessment visits.
  Data will be maintained on secure servers behind the firewalls at the two study sites: Kaiser Permanente Washington (KPWA) and the University of California, San Francisco (UCSF). De-identified or limited datasets containing individual-level data on which publications are based will be made available to qualified researchers for specified analyses. We will make the data available to users only under a data-use agreement (DUA).
Supporting Information: Study Protocol, SAP
Time Frame: Data can be requested after the primary study paper is accepted for publication, up until 5 years after study completion.
Access Criteria: Individuals interested in using KPWA data will be required to complete a standard form, sign a Data Use Agreement (DUA) and provide documentation of IRB approval. Data may then be accessed by qualified researchers via KPWA's Secure File Transfer (SFT) site. User registration will be required in order to access or download data files. As part of the registration process, users must agree to the conditions of use governing access to the data, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data resource.

REFERENCES:
- [Background] Lee SJ, Larson EB, Dublin S, Walker R, Marcum Z, Barnes D. A Cohort Study of Healthcare Utilization in Older Adults with Undiagnosed Dementia. J Gen Intern Med. 2018 Jan;33(1):13-15. doi: 10.1007/s11606-017-4162-3. No abstract available. PMID 28849435
- [Background] Barnes DE, Zhou J, Walker RL, Larson EB, Lee SJ, Boscardin WJ, Marcum ZA, Dublin S. Development and Validation of eRADAR: A Tool Using EHR Data to Detect Unrecognized Dementia. J Am Geriatr Soc. 2020 Jan;68(1):103-111. doi: 10.1111/jgs.16182. Epub 2019 Oct 14. PMID 31612463
- [Background] Palazzo L, Hsu C, Barnes DE, Gray MF, Greenwood-Hickman MA, Larson EB, Dublin S. Patient and caregiver perspectives on a tool to increase recognition of undiagnosed dementia: a qualitative study. BMC Geriatr. 2021 Oct 26;21(1):604. doi: 10.1186/s12877-021-02523-0. PMID 34702167